CLINICAL TRIAL: NCT04288440
Title: Pathological Features of Epiretinal Membranes in Silicone Filled Eyes
Brief Title: Characters of Epiretinal Membranes in Patients With Previous Vitrectomy for Retinal Detachment
Acronym: RD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sharif Yousef El Emam, Lecturer of Ophthalmology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IAA; Faculty of medicine (Other: Tanta University)
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Rhegmatogenous Retinal Detachment of Both Eyes (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Surgical Procedures, Operative; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone filled eyes (Active Comparator): Eyes filled with silicone oil
  Interventions: Procedure: Surgery; Device: Vitrectomy machine
- Idiopathic ERM (Active Comparator): Eyes not filled with silicone oil
  Interventions: Procedure: Surgery; Device: Vitrectomy machine

INTERVENTIONS:
Procedure: Surgery — Removal of epiretinal membrane and ILM
  Other Names: Invasive procedure
Device: Vitrectomy machine — Pars plana vitrectomy

SUMMARY:
31 patients were included in the study,15 cases with ERM in silicone filled eyes and 16 eyes with idiopathic ERM

DETAILED DESCRIPTION:
This is a prospective study that included 31 patients and was performed in Tanta University Eye Hospital in cooperation with the Pathology Department, Tanta University, between January 2018 and June 2019. The approval of the ethical committee of the Faculty of Medicine in Tanta University was obtained, and the study was conducted in accordance with the 1964 Helsinki Declaration and its later amendment. A detailed informed written consent was signed by all study participants. The research is not funded by the university or any organization or entity.

Fifteen cases had pars plana vitrectomy for rhegmatogenous retinal detachment nine months earlier with ERM detected by OCT one day before silicone oil removal. The other 16 cases matched for age and gender with idiopathic ERM and were included as a control. Histopathological features of the ERMs were compared between the two groups.

All patients have undergone complete ophthalmic evaluation including: best corrected visual acuity (BCVA) by Snellen chart that was converted to log MAR for statistical analysis, anterior segment examination by slit lamp, posterior segment examination by slit lamp bimicroscopy using +78 D lens and indirect Ophthalmoscopy, and Spectral domain optical coherence tomography (SD-OCT) (Spectralis; Heidelberg Engineering,Heidelberg, Germany) was performed for all patients before surgery.

The investigators excluded patients with previous intraocular surgery (except cataract surgery) for the control group, diabetes mellitus/diabetic retinopathy, coincident retinal pathology as choroidal neovascular membrane and age related macular degeneration, previous laser photocoagulation, intravitreal injection of Triamcinolone Acetonide or antivascular endothelial growth factor (anti-VEGF) agents, prior intra-ocular inflammation, retinal degenerations, neovascularization or rubeosis and vascular disorders e.g. retinal vein or artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Fifteen cases had pars plana vitrectomy for rhegmatogenous retinal detachment nine months earlier with ERM detected by OCT one day before silicone oil removal.
2. The other 16 cases matched for age and gender with idiopathic ERM and were included as a control. Histopathological features of the ERMs were compared between the two groups.

   -

Exclusion Criteria:the investigator excluded 1-patients with previous intraocular surgery (except cataract surgery) for the control group.

2- Diabetes mellitus/diabetic retinopathy. 3-Coincident retinal pathology as choroidal neovascular membrane and age related macular degeneration.

4-previous laser photocoagulation, intravitreal injection of Triamcinolone Acetonide or antivascular endothelial growth factor (anti-VEGF) agents.

5- prior intra-ocular inflammation, retinal degenerations.

6-Neovascularization or rubeosis and vascular disorders e.g. retinal vein or artery occlusion.

-

Ages: 42 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of GFAP and CD cells in idiopathic and silicone oil ERM | 6 months
  Percentage of glial fibrillary acid protein positive cells and number of cluster of differentiation cells in idiopathic and silicone oil ERM

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Shafik, MD, Study Chair — Tanta University
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams GW, Azen SP, McCuen BW 2nd, Flynn HW Jr, Lai MY, Ryan SJ. Vitrectomy with silicone oil or long-acting gas in eyes with severe proliferative vitreoretinopathy: results of additional and long-term follow-up. Silicone Study report 11. Arch Ophthalmol. 1997 Mar;115(3):335-44. doi: 10.1001/archopht.1997.01100150337005. PMID 9076205
- See also: medical link that contains hundreds of scientific papers — https://www.ncbi.nlm.nih.gov.